CLINICAL TRIAL: NCT00912210
Title: Higher Protein Diet and Exercise for Optimal Weight Loss in Elderly Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Ellen Evans, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UIUC IRB 07782
Record Dates: First submitted 2009-05-29; First posted 2009-06-03 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-05

CONDITIONS: Bone and Body Composition; Obesity; Metabolic Syndrome; Physical Function; Quality of Life
MeSH Terms: conditions — Obesity; Metabolic Syndrome | interventions — Carbohydrates; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Higher protein (Active Comparator)
  Interventions: Dietary Supplement: Whey protein isolate
- Higher carbohydrate (Placebo Comparator)
  Interventions: Dietary Supplement: Maltodextrin powder supplement

INTERVENTIONS:
Dietary Supplement: Whey protein isolate — Loss of 10% baseline weight over 6 months, with whey protein isolate supplemented at 50g/day (two 25 g doses taken at breakfast and afternoon snack mixed with food or beverage)
  Arms: Higher protein
Dietary Supplement: Maltodextrin powder supplement — Loss of 10% baseline weight over 6 months, with whey protein isolate supplemented at 50 g / day (two 25 g doses at breakfast and afternoon snack mixed with food or beverage)
  Other Names: carbohydrate, starch
  Arms: Higher carbohydrate

SUMMARY:
The broad aim is to determine efficacy of a weight loss diet higher in protein and lower in carbohydrate combined with low intensity exercise to favorably impact body composition, bone health, physical function, metabolic disease and quality of life compared to a conventional higher carbohydrate diet in overweight women over age 60.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index > 28 kg/m²
* Clearance of primary physician to participate in diet and mild exercise

Exclusion Criteria:

* Medical condition contraindicating prescribed diet and exercise regimen
* Type 2 Diabetes Mellitus
* Physically active lifestyle (>30 min moderate physical activity 2+ times weekly)

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-04

PRIMARY OUTCOMES:
Bone and body composition: Weight, percent fat, muscle and fat distribution in the thigh and abdomen and bone density and structural quality assessed by DXA and structural MRI | Baseline and post 6 months weight loss

SECONDARY OUTCOMES:
Physical function: balance, gait, strength and activities of daily living | Baseline and post 6 months weight loss
Quality of life | Baseline and post 6 months weight loss
Metabolic syndrome: insulin resistance, blood pressure, blood lipids, waist circumference | Baseline and post 6 months weight loss
Acid-base balance | Baseline and post 1 and 6 months weight loss

CONTACTS AND LOCATIONS:
Overall Officials: Ellen M Evans, PhD, Principal Investigator — University of Illinois at Urbana-Champaign; Donald K Layman, PhD, Principal Investigator — University of Illinois at Urbana-Champaign; Edward McAuley, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States